CLINICAL TRIAL: NCT00924300
Title: Magnetoencephalography (MEG) and Magnetic Resonance Imaging (MRI) Studies of Typical and Atypical Cognitive Processes in Children and Adolescents
Brief Title: Study to Test the Usefulness of Magnetoencephalography (MEG) Imaging of Cognition in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0217-09-FB
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Cognition
Keywords: feasibility of MEG in pediatric populations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: children and/or adolescents with psychiatric disorder
- controls: typically-developing children/adolescents

SUMMARY:
The primary objective of this protocol is to test the feasibility and utility of obtaining magnetoencephalography (MEG) recordings in healthy children and also in children who have a psychiatric or developmental disorder. Secondary objectives are to examine and compare typical and atypical motor, sensory, and cognitive functioning as recorded by MEG, and to identify subpopulation groups for which MEG may be optimal in order to establish feasibility of future hypothesis-driven MEG research.

DETAILED DESCRIPTION:
Healthy children and those who have a psychiatric or developmental disorder will undergo MEG recording to evaluate whether such children are candidate MEG subjects. Essentially, this feasibility study will examine whether children can remain still enough, complete simple tasks, and produce neurophysiologically consistent responses that would warrant full size studies.

ELIGIBILITY:
Inclusion Criteria:

* May or may not have a psychiatric or developmental disorder diagnosis.
* Outpatient at study entry.
* Age 4-18 (inclusive).
* Male or female.
* Have ability to sit still for 5 minutes or longer.
* Have ability to comply with basic instructions.
* Provide written informed assent if willing and able, per local IRB requirements before any study specific procedures are performed.
* Parent or legal guardian provide written informed consent before any study specific procedures are performed.

Exclusion Criteria:

* Ferrous metal permanently attached on or implanted in their body.
* Metal braces on teeth (i.e. Invisalign braces and cavity fillings are permitted).
* Has major medical condition, including cancer or hepatitis.
* Has confounding multiple psychiatric and/or developmental diagnoses, as judged by the principal or co-investigator.
* Known history or diagnosis of alcohol or substance abuse/dependence.
* Unable or unwilling to comply with the protocol.
* Anyone deemed as not appropriate for study participation, as deemed by the principal investigator.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children and adolescents with or without a psychiatric disorder
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-07-15 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Magnetoencephalography (MEG) activation | 2-4 hour single visit
  Task assignment is not randomized, but will be selected based upon age, developmental level of abilities, and disorder of interest, resulting in subjects and subgroups completing different tasks chosen by the principal investigator. Tasks include: auditory stimulation, visual stimulation, somatosensory stimulation, motor tasks, and baseline brain function. While the assigned tasks are performed, the MEG will silently record neuromagnetic responses on a 306-channel whole head Vector View system.

CONTACTS AND LOCATIONS:
Overall Officials: Tony W Wilson, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States